CLINICAL TRIAL: NCT03196115
Title: Biomarker for Hyaline Fibromatosis Syndrome - An International, Multicenter, Epidemiological Protocol
Brief Title: Biomarker for Hyaline Fibromatosis Syndrome (BioHFS)
Acronym: BioHFS
Status: Withdrawn | Type: Observational
Why Stopped: Transition to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BHFS 06-2018
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Hyalinosis; Hyaline Membrane Disease; Juvenile Hyaline Fibromatosis; Fibromatosis Hyalinica Multiplex Juvenilis; Skin and Connective Tissue Diseases
Keywords: Hyaline Fibromatosis Syndrome; Biomarker
MeSH Terms: conditions — Hyaline Membrane Disease; Hyaline Fibromatosis Syndrome; Skin and Connective Tissue Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of Mass-spectometry, a blood sample will be taken from patient via using a dry blood spot filter card. To proof the correct Hyaline fibromatosis syndrome diagnosis in those patients where up to the enrolment in the study no genetic testing has been done, sequencing of Hyaline fibromatosis syndrome will be done.
  The analyses will be done at:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observation: Patients with Hyaline fibromatosis syndrome or high-grade suspicion for Hyaline fibromatosis syndrome

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Hyaline fibromatosis syndrome from the blood

DETAILED DESCRIPTION:
Hyaline fibromatosis syndrome (HFS) is rare autosomal recessive disease characterized by the deposition of amorphous hyaline material in skin and visceral organs. It represents a disease spectrum with infantile systemic hyalinosis (ISH) being the severe form and juvenile hyaline fibromatosis (JHF) being the mild form. Dermatologic manifestations include thickened skin, perianal nodules, and facial papules, gingival hyperplasia, large subcutaneous tumors on the scalp, hyperpigmented plaques over the metacarpophalangeal joints and malleoli, and joint contractures. ISH shows a severe visceral involvement, recurrent infections, and early death.

The lesions appear as pearly papules or fleshy nodules. The severity is variable. Some individuals present in infancy and have additional visceral or systemic involvement, which can lead to early death. These patients may show intractable diarrhea and increased susceptibility to infection. Other patients have later onset of a milder disorder affecting only the face and digits. Additional features include gingival hypertrophy, progressive joint contractures resulting in severe limitation of mobility, osteopenia, and osteoporosis. Histologic analysis of skin lesions shows proliferation of spindle-shaped cells forming strands in a homogeneous and hyaline eosinophilic extracellular material in the dermis.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

Therefore it is the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent will be obtained from the parents before any study related procedures.
* Patients of both gender older than 2 months
* The patient has a diagnosis of Hyaline fibromatosis syndrome or a high-grade suspicion for Hyaline fibromatosis syndrome

High-grade suspicion present, if one or more inclusion criteria are valid:

* Positive family anamnesis for Hyaline fibromatosis syndrome
* Coarse facies
* Subcutaneous nodule
* Gingival fibromatosis
* Skeletal muscle atrophy
* Progressive flexion contractures

Exclusion Criteria:

* No Informed consent from the parents before any study related procedures.
* Patients of both gender younger than 2 months
* No diagnosis of Hyaline fibromatosis syndrome or no valid criteria for profound suspicion of Hyaline fibromatosis syndrome

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Hyaline fibromatosis syndrome or high-grade suspicion for Hyaline fibromatosis syndrome
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Sequencing of the Hyaline Fibromatosis Syndrome related gene | 4 weeks
  Next-Generation Sequencing (NGS) of the ANTXR2 gene will be performed. The mutation will be confirmed by Sanger sequencing.

SECONDARY OUTCOMES:
The Hyaline Fibromatosis Syndrome specific biomarker candidates finding | 24 months
  The quantitative determination of small molecules (molecular weight 150-700 kD, given as ng/μl) within a dried blood spot sample will be validated via liquid chromatography multiple reaction-monitoring mass spectrometry (LC/MRM-MS) and compared with a merged control cohort. The statistically best validated molecule will be considered as a disease specific biomarker.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (3):
- Centogene AG, Rostock, Germany
- NIRMAN Navi Mumbai Institute of Research In Mental And Neurological Handicap/Pediatric Geneticist, Mumbai, India
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: Undecided